CLINICAL TRIAL: NCT04764214
Title: An Open-label, Single-Arm, Phase 2 Trial of Stereotactic Radiotherapy for Patients With Residual Oligometastases of NSCLC After 3rd Generation EGFR-TKIs
Brief Title: SRT for Residual Oligometastases of NSCLC After 3rd Generation EGFR-TKIs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-NSCLCSBRT-1
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: NSCLC Stage IV; EGFR Activating Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3rd generation EGFR-TKI+ SRT (Experimental): Patients were treated with the intent to ablate all residual disease with consolidative SRT. EGFR-TKI treatment was continued during and after consolidative SRT until disease progression or intolerable toxicity.
  Interventions: Drug: 3rd generation EGFR-TKI; Radiation: Consolidative SRT

INTERVENTIONS:
Drug: 3rd generation EGFR-TKI — Osimertinib will be administered orally at the dose of 80 mg once daily.
  Other Names: Osimertinib
Radiation: Consolidative SRT — Patients who possess oligoresidual disease after 3rd generation EGFR-TKI therapy will be treated with the intent to ablate all residual disease with consolidative SRT. The choice of dose-fractionation regimen is at the discretion of the treating radiation oncologist. TKI will be continued during and after consolidative SRT until disease progression or intolerable toxicity.

SUMMARY:
This study is an open-label, single-arm phase 2 trial to evaluate the efficacy and safety of stereotactic radiotherapy (SRT) for patients with oligo-residual NSCLC after 3rd generation EGFR-TKIs.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosis of pathologically confirmed NSCLC by tumor biopsy and/or fine-needle aspiration.
* The patient has a diagnosis of American Joint Committee on Cancer (AJCC) 8th Edition stage IV NSCLC.
* The patient receives 3rd generation EGFR-TKI in the first line setting.
* The patient is ≥18 years of age and ≤75 years of age at the time of screening.
* The patient's Karnofsky performance score (KPS) is ≥70 at study entry.
* The patient has adequate baseline tumor assessment before initiation of 3rd generation EGFR-TKI.
* The patient has at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
* The patient presents with a residual "oligometastatic" state after 3rd generation EGFR-TKI therapy that would be amenable to consolidative SRT in the opinion of the investigator.
* The patient has signed informed consent.
* EGFR Exon19 deletion or Exon21 L858R mutation

Exclusion Criteria:

* History of another malignancy or concurrent malignancy. Patients with cervical carcinoma in situ or adequately treated basal cell carcinoma who have been disease free for > 5 years are eligible.
* The patient is pregnant (confirmed by serum b-HCG if applicable) or is breastfeeding.
* Patients with uncontrolled epilepsy, mental disorders, drug abuse, or social condition that may affect compliance or ability to sign a written informed consent in the opinion of the investigator.
* Patients with residual metastatic disease after 3rd generation EGFR-TKI therapy that is deemed not amenable to consolidative SRT.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | Two years
  PFS was measured from the date of enrollment to the date of disease progression as defined by Response Evaluation Criteria in Solid Tumor (RECIST) Version 1.1 or death due to any cause, whichever occurred first. For patients whose disease did not progress, PFS was evaluated by censoring patients at their most recent imaging.

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | Two years
  Treatment-related adverse events were assessed and graded according to CTCAE v. 5.0.
Overall Survival | Two years
  OS was defined as the time from the date of enrollment until death by any cause. Participants still alive at the time of data analysis were censored at the date of last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Zhengfei Zhu, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Zhou Y, Peng L, Liang F, Chu L, Chu X, Yang X, Zhang J, Guo T, Jiang S, Pang Y, Wang Z, Zhang L, Ni J, Zhu Z. Safety and efficacy of consolidative stereotactic radiotherapy for oligo-residual EGFR-mutant non-small cell lung cancer after first-line third-generation EGFR-tyrosine kinase inhibitors: a single-arm, phase 2 trial. EClinicalMedicine. 2024 Sep 26;76:102853. doi: 10.1016/j.eclinm.2024.102853. eCollection 2024 Oct. PMID 39398493